CLINICAL TRIAL: NCT05101551
Title: A Phase I Protocol for Relapsed Pediatric AML to Determine the Safety and Efficacy of the PARP Inhibitor Talazoparib in Combination With Chemotherapy
Brief Title: Study of Talazoparib in Combination With Chemotherapy in Relapsed Pediatric AML to Determine Safety and Efficacy
Acronym: PARPAML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Norman J. Lacayo (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Norman J. Lacayo, Instructor Pediatrics - Hematology/Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-66573; PEDSHEMAML0008 (Other: OnCore); POE22-01 (Other: POETIC study number); Pro00060706 (Other: Advarra IRB number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: PARP Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — talazoparib; Topotecan; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talazoparib with topotecan and gemcitabine (Experimental): Talazoparib will be administered orally on Days 1 to 5 concurrently with topotecan and a single dose of gemcitabine on Day 1 of 28 day cycle for 1 or 2 cycles. Subjects on dose level 5 will receive an additional 5 day treatment course of talazoparib on days 15-19.
  Interventions: Drug: Talazoparib; Drug: Topotecan; Drug: Gemcitabine

INTERVENTIONS:
Drug: Talazoparib — Talazoparib will be administered in escalating doses based on current dose level.
  * Dose Level 1: 400 µg/m2/dose once daily
  * Dose Level 2: 600 µg/m2/dose BID on Day 1, then daily on Days 2 to 5
  * Dose Level 3: 600 µg/m2/dose BID on Day 1, then daily on Days 2 to 5
  * Dose Level 4: 600 µg/m2/dose BID on Day 1, then daily on Days 2 to 5
  * Dose Level 5: 600 ug/m2/dose BID on Day 1, then daily on Days 2 to 5 and 15 to19
  Other Names: Talzenna
Drug: Topotecan — Administered IV route on Days 1 to 5
  * Dose Level -2: 1 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level -1: 2 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level 1: 2 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level 2: 2 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level 3: 3 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level 4: 4 mg/m2/dose once daily by IV days 1 to 5
  * Dose Level 5: 4 mg/m2/dose once daily by IV days 1 to 5
  Other Names: Hycamtin
Drug: Gemcitabine — Single dose (IV) of gemcitabine on Day 1 of each 28 day cycle for 1 cycle.
  * Dose Level -2: 600 mg/m2/dose once daily by IV days 1
  * Dose Level -1: 600 mg/m2/dose once daily by IV days 1
  * Dose Level 1: 1200 mg/m2/dose once daily by IV days 1
  * Dose Level 2: 1200 mg/m2/dose once daily by IV days 1
  * Dose Level 3: 1200 mg/m2/dose once daily by IV days 1
  * Dose Level 4: 1200 mg/m2/dose once daily by IV days 1
  * Dose Level 5: 1200 mg/m2/dose once daily by IV days 1
  Other Names: Gemzar; Infugem

SUMMARY:
This is a Phase 1, open label, multicenter, dose finding study with dose expansion intended to evaluate the safety and tolerability of talazoparib in combination with conventional chemotherapy. Preliminary estimates of efficacy will be obtain through a dose expansion cohort receiving the maximum tolerated dose from the dose escalation phase of the study.

This study aims to determine the safety of talazoparib in combination with conventional chemotherapy and to establish the maximum tolerated dose of all 3 drugs when given in combination. A preliminary estimate of efficacy through a dose expansion phase is a secondary aim.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≤ 21 years.
2. Acute myeloid leukemia (AML) OR acute leukemia of ambiguous lineage (acute undifferentiated leukemia or mixed phenotype acute leukemia), specified as either refractory (persistent leukemia after at least 2 courses of induction chemotherapy) or relapsed, and further defined as any one of the criteria below:

   1. Bone marrow specimen ≥ 5% leukemic blasts by flow, as assessed by Hematologics Inc.
   2. A single bone marrow specimen with at least 2 tests demonstrates ≥ 1% leukemic blasts by flow cytometry (as assessed by Hematologics Inc), AND at least one of the following:

      * Karyotypic abnormality with at least 1 metaphase similar or identical to diagnosis
      * FISH abnormality identical to one present at diagnosis
      * PCR or NGS-based demonstration of leukemogenic lesion identical to diagnosis
   3. Rising MRD > 0.1% by flow cytometry on ≥ 2 serial samples, as assessed by Hematologics Inc.
   4. If an adequate bone marrow sample is not obtained, subjects may be enrolled if there is unequivocal evidence of leukemia based on ≥ 5% blasts in the peripheral blood
3. > 60 days has passed since hematopoietic stem cell transplant.
4. Patients who have undergone previous allogeneic stem cell transplantation who are otherwise eligible must also be without evidence of any active graft versus host disease (GVHD), and off calcineurin inhibitors for at least 28 days (four weeks) prior to therapy. A physiologic dose of prednisone up to 3 mg/m2 (and a maximum of 7.5 mg) or equivalent other steroid dose is allowable.
5. A minimum of 14 days has passed since completion of myelosuppressive therapy or gemtuzumab ozogamicin and all nonhematologic toxicities have resolved to Grade 0 or 1.
6. A minimum of 24 hours has elapsed since the patient has completed any low-dose or non-myelosuppressive therapy (e.g., hydroxyurea or low-dose cytarabine (up to 100 mg/m2).
7. Lansky (subjects ≤ 16 years old) or Karnofsky (subjects > 16 years old) score ≥ 50.
8. WBC ≤ 50,000/uL. This may be achieved using cytoreductive therapy such as hydroxyurea or low-dose cytarabine (up to 100 mg/m2/dose)
9. Total bilirubin ≤ 2.0 x institutional upper limit of normal (ULN) for age.
10. AST/ALT ≤ 5 x ULN for age
11. Left ventricular ejection fraction ≥ 40% or ECHO shortening fraction ≥ 25%.
12. Estimated serum creatinine ≥ 60 mL/min/1.73m2

Exclusion Criteria:

1. Patients receiving or planning to receive ANY concurrent cancer therapy, including chemotherapy, radiation therapy, immunotherapy or biologic therapy.
2. Patients with down syndrome.
3. Patients with Acute Promyelocytic leukemia (APL) or Juvenile Myelomonocytic Leukemia (JMML).
4. Patients with Bone Marrow Failure Syndrome.
5. Pregnant subjects or those unwilling to use an effective method of birth control.
6. Female subjects with infants who do NOT agree to abstain from breastfeeding.
7. Inability or unwillingness of legal guardian/representative to give written informed consent.
8. Patients with uncontrolled systemic fungal, bacterial, viral or other infection.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT). | 28 days after starting therapy (ie, single course of therapy).
  Patient safety is assessed as dose limiting toxicity (DLT). The outcome is the number of DLT events. A DLT event is defined as:
  * Hematologic DLT - Failure to recover peripheral ANC to > 200/µL or non-transfusion-dependent platelets to > 20,000/µL by Day 43 from the start of Cycle 1 of chemotherapy will be considered a DLT, unless the delay in count recovery is due to another identifiable factor
  * Non-Hematologic DLT-Any ≥ Grade 4 non-hematological organ toxicity, including Hy's Law case is a DLT with the following exceptions:
  * Grade 4 infection or fever ≤ 7 days in duration.
  * Grade 4 electrolyte or laboratory abnormalities correctable with supportive therapy or that resolve to < Grade 3 within 72 hours.
  * Grade 4 elevation in hepatic transaminases that resolves to ≤ Grade 2 within 7 days.
  * Grade 4 tumor lysis syndrome must resolve in ≤ 7 days without evidence of end-organ damage.

SECONDARY OUTCOMES:
Objective Response (OR) | 28 days
  Objective response includes all participants that achieve complete or partial response, and assessed for all participants treated at the maximum tolerated dose.
  * Complete remission: Bone marrow MRD < 5% by flow cytometry, ANC ≥ 500/μL AND platelets ≥ 50,000/μL,without transfusions,No extramedullary disease
  * Complete remission without hematologic recovery: Bone marrow MRD < 5% by flow cytometry, One of ANC ≥ 500/μL OR platelets ≥ 50,000/μL,without transfusions, No extramedullary disease
  * Partial response: Decrease of at least 50% of blasts by MRD and ≥ 5% to 25% blasts by flow cytometry.Enrolled patients with fewer than 5% blasts by MRD are not evaluable for PR.
  * No response: No change in clinical or laboratory status.For patients with < 5% of blasts at enrollment, no response is defined as failure to achieve MRD negative CR or MRD negative CRi.
  * Progressive Disease: Deterioration of initial disease status
  * MRD negative: < 0.05% of leukemic blasts by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Lacayo, MD, Principal Investigator — Stanford Universiy
Locations (9):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Stanford University, Stanford, California
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pennsylvania State University Hershey Medical Center, Hershey, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No